CLINICAL TRIAL: NCT06383299
Title: Turkish Validity and Reliability of Calgary Sleep Apnea Quality of Life Index
Brief Title: The Validity and Reliability Study of Turkish Version of Calgary Sleep Apnea Quality of Life Index
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Bahar Anaforoglu, assoc.prof, Ankara Yildirim Beyazıt University
Other Study IDs: AnkaraYbuMNC
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Obstruvtive Sleep Apnea Syndrome (OSAS)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: untreated group
- 2: cpap treatment group

SUMMARY:
The aim of this study is to investigate its validity and reliability of the questionarre whose original English name was "Calgary Sleep Apnea Quality of Life Index" which we plan to translate into Turkish as Sleep Apnea Quality of Life Index.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Apnea hypopnea index (AHI) of ≥5

Exclusion Criteria:

* Presence of sleep disturbances other than OSAS
* Presence of active alcohol or drug addiction
* Psychiatric impairment
* Cognitive impairment
* Recent acute illness (such as myocardial infarction) that may adversely affect their quality of life
* Difficulty in communicating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obstructive sleep apnea syndrome
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Calgary Sleep Apnea Quality of Life İndex (C-SAQLI) | time 0 and two week later
  The C-SAQLI was developed as a sleep apnea specific quality of life instrument It is a 35-item questionnaire that measures the negative impact of sleep apnea on daily functions, social interactions, emotional functions, and symptoms. Items are scored on a 7-point scale with "all of the time" and "not at all" being the most extreme responses. Item and domain scores are averaged to yield a composite total score between 1 and 7. Higher scores represent better quality of life.
Short Form 36 | time 0 and two week later
  The SF-36 is a multipurpose self-administered health survey consisting of 36 questions divided into 8 individual domains. These 8 sections are as follows; (1) physical functioning , (2) role physical , (3) bodily pain, (4) general health perceptions; (5) vitality , (6) social functioning, (7) role emotional, and (8) general mental health.
Epworth Sleepiness Scale | time 0 and two week later
  The ESS is an eight-item questionnaire that measure daytime sleepiness. The questionnaire is in a four-Likert (0-3) response format and the score ranges from 0 to 24. Higher scores indicate more daytime sleepiness.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yildirim Beyazıt University, Ankara, Turkey (Türkiye)